CLINICAL TRIAL: NCT03732313
Title: Altering Toenail Biomechanic in Managing Ingrown Toenail.Randomized Clinical Trial.
Brief Title: Altering Toenail Biomechanic in Managing Ingrown Toenail.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, Assistant professour general surgery zagazig university Egypt, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27908201300677
Record Dates: First submitted 2018-10-27; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Ingrown Toenail
Keywords: Ingrown toenail; Biomechanic; Central resection; Recurrence
MeSH Terms: conditions — Nails, Ingrown; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Central toenail resection (Active Comparator): Under local ring anaesthesua using xylocaine injection in base of big toe ,Surgical resection of the central part of toenail with underlying germinal matrix.the defect is sutures by prolene.
  Interventions: Procedure: Central toenail resection
- wedge toenail resection (Active Comparator): Under local ring anaesthesiausing xylocaine injection around the base of big toe. Resect lateral wedge of toenail with removal of ingrown toenail and periungual skin. The wound is then sutured.
  Interventions: Procedure: Wedge toenail resection

INTERVENTIONS:
Procedure: Central toenail resection — Using local aneasthesia, resection of central part of toenail with germinal matrix.
  Other Names: Surgical resection
  Arms: Central toenail resection
Procedure: Wedge toenail resection — Using local anaesthesia,we remove lateral part of toenail .
  Other Names: Surgical resection
  Arms: wedge toenail resection

SUMMARY:
Ingrown toenail is commonly met in clinical practice.treatment may be non-operative and operative treatment.operative trestment depends on lateral wedge resection of the nail. The idea is to change toenail biomechanics by central toenail resection.

DETAILED DESCRIPTION:
The aim of this study is to compare between central toenail resection with ordinary lateral wedge resection in managing ingrown toenail. This study was performed on 100 patients divided into 2 groupd each is 50 patients. Group A underwent central resection while group B underwent lateral toenail resection.

ELIGIBILITY:
Inclusion Criteria:

* patient with ingrown toenail
* Patients from 10 years up to 35 years

Exclusion Criteria:

* patients with concurrent toe deformity
* patients less than 10 years or more than 35 years

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain on visual analog score for pain | six month
  All patients are pain free after 5 days postoperative
Intraoperative time measured in minutes | Six month
  All operations end within 15 minutes.

SECONDARY OUTCOMES:
Recurrence after operation | six month
  Recurrence is followed up by asking the patient to follow up in outpatient clinic after six month and also,by calling the patients in telephone.

IPD SHARING:
Plan to Share IPD: No